CLINICAL TRIAL: NCT05143411
Title: Evaluation of a Mobile Application to Optimize Decision-making in Self-management and Reduction of Complications in Persons With Type 1 Diabetes
Brief Title: Evaluation of a Mobile Application to Optimize Self-decision on Metabolic Control in Persons With Type 1 Diabetes
Acronym: DM-BLUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Iberoamericana (Other)
Collaborators: Clemson University (Other)
Responsible Party: Principal Investigator, Jenny Lujan Cepeda Marte, Doctor, Universidad Iberoamericana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-2019-3C1-044
Record Dates: First submitted 2021-11-08; First posted 2021-12-03 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes type 1; insulin bolus calculator; macronutrients
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Evaluation Studies as Topic

STUDY DESIGN:
Intervention Model Description: Evaluating pre-test and post-test (pre and post glucose levels)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of mobile application (Experimental): Single arm: At the first time, the researcher will collect all glycemic levels before using the mobile application. Then, all the participants will receive the mobile application to select their main meals, breakfast, lunch, and dinner. Then, the application must calculate the insulin bolus according to their initial profile and the food before being eaten.
  Interventions: Other: PRE-test

INTERVENTIONS:
Other: PRE-test — we are going to verify glucose levels before (pre) and after (post) the use of the mobile application.
  Other Names: Post-Test

SUMMARY:
Adolescents with type 1 diabetes mellitus (T1 DM) tend to have poor metabolic control. There are no mobile applications in our language in our environment, and patients are accessible in addition to the difficulties involved in these manual calculations. One way to bridge the knowledge gaps in T1 DM self-management is by using technology to optimize metabolic control and reduce the risks of associated comorbidities, with a mobile application that helps optimize decision-making in self-management. This research aims to help people with type 1 diabetes to change the glycemic blood levels and to be able to calculate the food together with the amount of insulin with food from the region. To evaluate the acceptability and effectiveness of the application, the investigators will carry out a pilot evaluation test. The participants in this pilot test will be 20 people between 14 and 18 years old with T1DM, users of the pediatric diabetology service of the National Institute of Diabetes, Endocrinology, and Nutrition (INDEN).

DETAILED DESCRIPTION:
Metabolic lack of control in patients with type 1 diabetes Mellitus (T1DM) leads to kidney failure, non-traumatic amputations, blindness, and reduced life expectancy. In addition, determining the content of macronutrients in food is not the domain of many patients, particularly adolescents, or some physicians, making insulin adjustment difficult, one of the main failures of optimal metabolic control. One way to bridge the knowledge gaps in T1D self-management is by using technology to optimize metabolic control and reduce the risks of associated comorbidities, with a mobile application that helps optimize decision-making in self-management. And a reduction of complications in adolescents (14-18 years) with T1DM. This project aims to develop this application that contributes to decision-making and the reduction of comorbidities of adolescents with T1DM, following the policies of the Dominican state through Digital systems, together with its educational mission, technological access, and national competitiveness.

There are no mobile applications in use in the Dominican Republic for the self-management of chronic diseases. Therefore, the investigators have designed a mobile application with a postprandial insulin bolus calculator. In addition, the developers has added a list of foods from the region where users can select their foods and adjust them with the amount of insulin to metabolize them. The methodology includes a mixed approach (qualitative and quantitative) before starting the study and after three months of using the application.

To evaluate the acceptability and effectiveness of the application, we will carry out a pilot evaluation test. The participants in this pilot test will be 20 people between 14 and 18 years old with T1DM, users of INDEN. This experimental study has a systematized probabilistic sample from the center's master list. They were randomized, not controlled. Therefore, the participants are users of the pediatric diabetology service, and included prior explanation and approval of informed consent. These 20 participants will be recruited, ensuring the equitable distribution between gender and sociodemographic data of the mentioned group while maintaining the intention to treat.

Inclusion criteria:

-Patients between 14-18 years old with diabetes type 1.

Exclusion criteria

* Patients with Glomerular filtration rate less than 60 mL/min
* Inability to use electronic devices.
* Admission due to acute decompensation of T1DM in previous 3 months, presence of more than one severe monthly hypoglycemia, or any other circumstance that requires frequent visits and intensive care.
* Inability to sign the informed consent.

The investigators invited the participants to select foods and routinely use the mobile app's insulin bolus calculator for three months.

For data analysis, the researchers are going to perform the normality test for numerical variables. Then, the categorical data presentation will be with frequencies and percentages tables and the quantitative data as means and standard deviation, and use a non-Gaussian distribution, Kruskal-Wallis and Mann-Whitney tests.

The primary endpoint, HbA1c at the beginning of the study and the end of the third month of use of the application, will be analyzed with Kruskal-Wallis and Mann-Whitney tests and for pre-test and post-test comparisons of the study group, and the multifactorial analysis of variance (ANCOVA), baseline HbA1c level and at 3 months after using the application, taking into account age as covariates. The investigators are going to use for statistical analysis the Statistical Package for the Social Sciences (SPSS), and Excel of the data obtained.

ELIGIBILITY:
Inclusion Criteria:

* Persons with diabetes type 1

Exclusion Criteria:

* Persons with oral diabetes treatment.
* Glomerular filtration rate less than 60 mL/min

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Change in glucose levels | Day 01, Month 01
  We expect to find changes in glucose levels before each main meal

SECONDARY OUTCOMES:
Change in glycemic variability | Day 01, month 3
  we expect to find changes in variations of coefficients

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Iberoamericana, Santo Domingo, Nacional, Dominican Republic

IPD SHARING:
Plan to Share IPD: Yes
We will be presenting the results at the congress of the American Diabetes Association if it is accepted.
Supporting Information: Study Protocol, SAP
Time Frame: Starting six month after publication 2022
Access Criteria: It will be able on-demand, email to principal investigator at Iberoamerican University (UNIBE): j.cepeda1@unibe.edu.do
URL: http://www.unibe.edu.do

REFERENCES:
- [Background] Ewers B, Vilsboll T, Andersen HU, Bruun JM. The dietary education trial in carbohydrate counting (DIET-CARB Study): study protocol for a randomised, parallel, open-label, intervention study comparing different approaches to dietary self-management in patients with type 1 diabetes. BMJ Open. 2019 Sep 3;9(9):e029859. doi: 10.1136/bmjopen-2019-029859. PMID 31481560
- [Background] Darby A, Strum MW, Holmes E, Gatwood J. A Review of Nutritional Tracking Mobile Applications for Diabetes Patient Use. Diabetes Technol Ther. 2016 Mar;18(3):200-12. doi: 10.1089/dia.2015.0299. Epub 2016 Mar 7. PMID 26950679
- [Background] Goksen D, Atik Altinok Y, Ozen S, Demir G, Darcan S. Effects of carbohydrate counting method on metabolic control in children with type 1 diabetes mellitus. J Clin Res Pediatr Endocrinol. 2014;6(2):74-8. doi: 10.4274/Jcrpe.1191. PMID 24932599
- [Background] Dias VM, Pandini JA, Nunes RR, Sperandei SL, Portella ES, Cobas RA, Gomes MB. Effect of the carbohydrate counting method on glycemic control in patients with type 1 diabetes. Diabetol Metab Syndr. 2010 Aug 17;2:54. doi: 10.1186/1758-5996-2-54. PMID 20716374
- [Background] Son O, Efe B, Son NE, Akalin A, Kebapci N. Investigation on carbohydrate counting method in type 1 diabetic patients. Biomed Res Int. 2014;2014:176564. doi: 10.1155/2014/176564. Epub 2014 Aug 17. PMID 25202704